CLINICAL TRIAL: NCT04903301
Title: Patient Satisfaction With Contoura Vision Topography-Guided LASIK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rush Eye Associates (Other)
Responsible Party: Principal Investigator, Sloan W. Rush, MD, Principal Investigator, Rush Eye Associates
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CV-LASIK
Record Dates: First submitted 2021-05-21; First posted 2021-05-26 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Study Group (Experimental): Contoura Vision LASIK using Phorcides Analytic Software
  Interventions: Procedure: Contoura Vision LASIK

INTERVENTIONS:
Procedure: Contoura Vision LASIK — Topography-Guided LASIK using Phorcides Analytic Software

SUMMARY:
To evaluate patient reported outcomes associated with quality of vision before and after treatment with Contoura Vision Topography-Guided LASIK.

ELIGIBILITY:
Eligibility criteria: The study enrollment will include all willing patients with: pre-operative BCVA 20/20 for each eye individually, myopic refractive error up to -8.00 diopters, refractive astigmatism that ranges from 0 to 3 diopters, maximum spherical equivalent of -9.00 diopters, the designated age requirements, and only patients that have signed the informed consent document.

Exclusion criteria: Patients are excluded that are not willing to participate in a research trial, are unable to cooperate well enough to safely perform the procedure, fail to meet inclusion criteria, have ocular disease (including but not limited to keratoconus, macular degeneration, glaucoma, corneal dystrophy, dry eye syndrome and corneal scarring), and patients that have had previous ocular surgery. Any patients with known allergies to the post-operative medications or preservatives in the medications will also be excluded.

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-01 (Actual)

PRIMARY OUTCOMES:
Global Vision Satisfaction Index | 26 weeks
  Analog Score from Adapted from PROWL Survey

SECONDARY OUTCOMES:
Vision | 26 weeks
  Uncorrected Visual Acuity using ETDRS
Objective Scatter Index | 26 weeks
  HD Analyzer
Higher Order Corneal Aberrations | 26 weeks
  Galilei Topography

CONTACTS AND LOCATIONS:
Locations (1):
- Rush Eye Associates, Amarillo, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided